CLINICAL TRIAL: NCT06031675
Title: The αKlotho Protein-mediated NLRP3/Caspase-1/GSDMD Pathway Counteracts Myocardial Stunning: a Novel Mechanism for Exercise to Delay Cardiac Aging
Brief Title: Mechanism for Exercise to Delay Cardiac Aging
Status: Completed | Type: Observational
Sponsor: Xiao-dong Zhuang (Other)
Responsible Party: Sponsor-Investigator, Xiao-dong Zhuang, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: K0001
Record Dates: First submitted 2023-08-31; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Activity, Motor; Health Behavior
Keywords: vigorous intermittent lifestyle physical activity; wearable device; isokinetic performance
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intervention group: The intervention measures encompass the implementation of simulated vigorous intermittent lifestyle physical activity for all participants. The specific exercise regimen involves performing rope jumping activities three times a day, with each session aimed at surpassing the exercise threshold (not conducted in a continuous manner), where the heart rate should exceed 160 beats per minute. This routine will be undertaken five times a week, continuously for a span of 8 weeks.
  Interventions: Other: Vigorous intermittent lifestyle physical activity

INTERVENTIONS:
Other: Vigorous intermittent lifestyle physical activity — The specific exercise regimen involves performing rope jumping activities three times a day, with each session aimed at surpassing the exercise threshold (not conducted in a continuous manner), where the heart rate should exceed 160 beats per minute. This routine will be undertaken five times a week, continuously for a span of 8 weeks.

SUMMARY:
The goal of this clinicaltrial is to assess and compare isokinetic performance, surface electromyography, laboratory parameters, and cardiorespiratory function both before and after engaging in vigorous intermittent lifestyle physical activity(VILPA) within a healthy population.

The main question it aims to answer is:

[1] Does VILPA yield effective outcomes?

Throughout the course of the trial, participants will engage in a simulated regimen of vigorous intermittent lifestyle physical activity for a duration of 8 weeks. The efficacy of the exercise protocol will be quantified and evaluated through the utilization of a wearable device.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Adults
2. No exercise habits (more than 3 months)

Exclusion Criteria:

1. Exercising ≥ 3 times per week;
2. the presence of chronic diseases, such as hypertension, hyperglycemic states, etc;
3. have conducted an exercise program in the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University students
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Isometric Strength Test | 15 minutes
  Isokinetic muscle strength testing with the Isomed 2000
Surface electromyography | 30 minutes
Exercise Flat Test | 30 minutes
  cardiopulmonary function

SECONDARY OUTCOMES:
Fasting glucose | 5 minutes
Blood lipid | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lizhen Liao, PhD, Study Director — Department of Health, Guangdong Pharmaceutical University
Locations (1):
- Guangdong Pharmaceutical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No